CLINICAL TRIAL: NCT04561739
Title: Paclitaxel-coated Balloon for the Treatment of De-novo Non-complex Coronary Artery Lesions: an Open-label, Multicentre, Randomised, Non-inferiority Trial
Brief Title: Paclitaxel-coated Balloon for Treatment of De-novo Non-complex Coronary Artery Lesions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, LingTao, Professor in Cardiology, Director of the department of Cardiology, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAGE-FREE 1
Record Dates: First submitted 2020-09-03; First posted 2020-09-24 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: De Novo Stenosis; Coronary Artery Disease
Keywords: drug-coated balloons; percutaneous coronary intervention; de novo stenosis; drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-coated balloon (Experimental)
  Interventions: Device: Paclitaxel coated balloon
- Drug-eluting stent (Active Comparator)
  Interventions: Device: Sirolimus eluting stents

INTERVENTIONS:
Device: Paclitaxel coated balloon — The Paclitaxel coated balloon is a paclitaxel-eluting rapid exchange balloon catheter for PTCA. Paclitaxel is the pharmacologically active substance for anti-neointima, whereas iopromide, a well-tolerated nonionic x-ray contrast agent, acts as a release-supporting additive.
  The active drug coating is located on the surface of the balloon, which contains 3 μg Paclitaxel per 1 mm2. The spray coating of the mixture of paclitaxel and iopromide of the Swide is via ultrasound, with the crystal size<2um.
  Arms: Drug-coated balloon
Device: Sirolimus eluting stents — The device has a backbone of L605 cobalt chromium. The stent has a open cell, in-phase, peak-to-valley design. The strut thickness is 86 μm and has a stent profile less than 1.12mm. The polymer coating of the stent is a styrene-butadiene block copolymer. The antiproliferative drug concentration is at 9 ug/mm, which 80% of the drug is released by 30 days.
  Arms: Drug-eluting stent

SUMMARY:
The introduction of Bare-metal stents (BMS) since 1986 has alleviated the limitations of plain old balloon angioplasty (POBA) related elastic recoil and flow-limiting dissections. Later on, higher restenosis rates due to exaggerated neointimal growth in BMS has led to the development of drug-eluting stents (DES), which elutes an antiproliferative drug to the vessel wall and reduce the restenosis rate. However, late stent thrombosis and restenosis, with a hazard of nearly 2% per year after implantation, remained a concern and motivated the development of drug-coated balloons (DCB).

The advantages of DCB are that leaving no metal in the blood vessel and respect the vessel anatomy.

Recently, studies with the strategy of DCB angioplasty with bailout stenting have demonstrated safety and efficacy for the small-vessel disease. In the BASKET-SMALL 2 trial, which compared SeQuent Please DCB with EES or Taxus DES in the vessels that have reference diameter<3mm, showed that at 12-month follow-up, DCB was non-inferior to DES (MACE [cardiac death, non-fatal myocardial infarction, and target-vessel revascularisation] rates: 8% vs. 9%).

Although some small-scale RCT using surrogate endpoints have reported that no significant difference in MLD or late lumen loss between the two groups in large vessels, up to now, there is no large-scale RCT comparing the clinical outcomes of DCB versus DES in large vessels with de novo lesions.

Therefore, the investigators hypothesized that in patients undergoing non-complex percutaneous coronary intervention (PCI) for de-novo stenoses, drug-coated balloon (DCB) is non-inferior to drug-eluting stents (DES).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an indication for PCI due to acute or chronic coronary syndrome
2. Patients with de-novo, non-complex lesion* and underwent successful pre-dilation**
3. Patients who are able to complete the follow-up and compliant to the prescribed medication

   * Non-complex PCI is defined as

1. Vessels treated<3; stents implanted<3; lesions treated<3 or Total stent length<60 mm 2. Bifurcation does not require 2 stents 3. Non left main lesion 4. Non venous or arterial graft lesion 5. Non chronic total occlusion lesion 6. Do not require the use of atherectomy device

**Successful pre-dilation is defined as fulfilling all the following criteria

1. Thrombolysis In Myocardial Infarction [TIMI] flow =3
2. Without dissections type D, E, and F
3. Residual stenoses <30% after balloon pre-dilation (visual).
4. Without serious complication requiring the termination of PCI

Exclusion Criteria:

1. Under the age of 18
2. Unable to give informed consent
3. The patient is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential according to local practice)
4. Known contraindication to medications such as Heparin, antiplatelet drugs, or contrast.
5. Currently participating in another trial and not yet at its primary endpoint
6. The concurrent medical condition with a life expectancy of less than 2 years
7. Previous intracranial hemorrhage
8. In-stent stenosis requiring revascularization (defined as stenosis≥50% by visual or positive functional assessments in any vessel)
9. Atrial fibrillation
10. Prior CABG
11. Cardiogenic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2272 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-05-05 (Estimated); Study Completion 2027-05-05 (Estimated)

PRIMARY OUTCOMES:
Device-oriented Composite Endpoint (DoCE) | 24 months
  DoCE is a composite clinical endpoint of Cardiac cause death, Target vessel myocardial infarction (TV-MI), and Clinically and physiologically indicated target lesion revascularization (CI-TLR).

SECONDARY OUTCOMES:
Device-oriented Composite Endpoint (DoCE) | 1, 12, 36, and 60 months
  Rates of the DoCE beside the time point of primary endpoint
Cardiac cause death | 1, 12, 24, 36, and 60 months
  Rates of individual components of the DoCE
Target vessel myocardial infarction (TV-MI) | 1, 12, 24, 36, and 60 months
  Rates of individual components of the DoCE
Clinically and physiologically indicated target lesion revascularization (CI-TLR) | 1, 12, 24, 36, and 60 months
  Rates of individual components of the DoCE
Patient-oriented composite endpoint (PoCE) | 1, 12, 24, 36, and 60 months
  Patient-oriented composite endpoint (PoCE) defined as all-cause death, any stroke, any MI, and any clinically and indicated revascularisation)
All-cause death | 1, 12, 24, 36, and 60 months
  individual components of PoCE
Any MI | 1, 12, 24, 36, and 60 months
  individual components of PoCE
Any stroke | 1, 12, 24, 36, and 60 months
  individual components of PoCE
Any revascularisation | 1, 12, 24, 36, and 60 months
  individual components of PoCE
Any clinically and physiologically indicated revascularisation | 1, 12, 24, 36, and 60 months
Target vessel failure (TVF) | 1, 12, 24, 36, and 60 months
  Target vessel failure, defined as cardiovascular death, TV MI and clinically-indicated target vessel revascularisation
Clinical and physiologically indicated target vessel revascularization | 1, 12, 24, 36, and 60 months
Net adverse clinical events (NACE) | 1, 12, 24, 36, and 60 months
  Net adverse clinical events (NACE), define as POCE or BARC type 3 or 5 bleeding events
BARC type 3 or 5 bleeding events | 1, 12, 24, 36, and 60 months
BARC defined type 2, 3 or 5 bleeding events | 1, 12, 24, 36, and 60 months
Definite/Probable Stent thrombosis rates | 1, 12, 24, 36, and 60 months
  According to ARC-II classification
Device success | 0 day (during index PCI)
  Device success is defined by the following: DCB: 1.Successful delivery within 120 seconds (DCB in vessel) of the DCB device at the intended target lesion; 2.DCB is successfully dilated for at least 30 seconds and the device system is successfully withdrawn; 3.After DCB dilation, the target vessel has no flow limiting dissection (type D, E and F); and the final in-lesion residual stenosis is less than 30% by core laboratory QCA (preferred methodology) or visual assessment; 4.No bailout procedure by stent; DES: 1.1. Successful delivery, balloon expansion, and deployment of the first assigned device, at the intended target lesion; 2.Successful withdrawal of the device delivery system; 3. 3. Attainment of a final in-stent residual stenosis of <20% by core laboratory QCA (preferred methodology) or visual assessment;
Procedure success during PCI | 7 days
  Device success + without the occurrence of DoCE + no stent thrombosis at discharge during the index procedure hospital stay (maximum of 7 days).
Clinically relevant ischemic or bleeding events | 1, 12, 24, 36, and 60 months
  Time from randomization to the occurrence of first any ischemic or bleeding endpoints, including all-cause death, any stroke, MI, BARC-defined type 3 bleeding, any revascularization and BARC-defined type 2 bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, M.D., Ph.D., Study Chair — Xijing Hospital; Patrick Serruys, M.D., Ph.D., Study Chair — National University of Ireland, Galway; Yoshinobu Onuma, M.D., Ph.D., Study Chair — National University of Ireland, Galway; Chao Gao, M.D., Ph.D., Study Chair — Xijing Hospital
Locations (1):
- Ling Tao, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang P, Zhou J, Gao H, Hu T, Sun D, Wang Q, Jiang H, Yin Z, Wen S, Jin Y, Chen H, Yuan M, Zhong L, Hu S, Lian Z, Jiang Z, Xia J, Liu J, Fu G, He X, Zhu B, Garg S, Onuma Y, Wang D, Serruys PW, Gao C, Tao L. Impact of sex on outcomes in patients treated with drug-coated balloons versus drug-eluting stents for de novo coronary artery lesions: Insights from the REC-CAGEFREE I trial. BMC Med. 2026 Jan 22. doi: 10.1186/s12916-026-04649-7. Online ahead of print. PMID 41572254
- [Derived] Bai X, Gao H, Lv Y, Sun D, Wang Q, Yin Z, Wen S, Jin Y, Chen H, Yuan M, Zhong L, Hu S, Lian Z, Zeng H, Pan H, Liu J, Fu G, Zhang R, He X, Capodanno D, Garg S, Onuma Y, Wang D, Serruys PW, Gao C, Tao L. Impact of Chronic Kidney Disease on Outcomes With Drug-Coated Balloons Versus Drug-Eluting Stents: Insights From the REC-CAGEFREE I Trial. Catheter Cardiovasc Interv. 2026 Jan;107(1):304-314. doi: 10.1002/ccd.70348. Epub 2025 Nov 20. PMID 41264778
- [Derived] Tao L, He X, Shen G, Wu M, He Y, Ma L, Yang F, Ji Z, Wang H, Wu Y, Fang Z, Jiang H, Wen S, Jin Y, Chen H, Zhong L, Hu S, Liu Y, Li F, Zhou J, Ouyang F, Zhang Z, Zhu B, Zhang R, Fu G, Liu J, Jiang Z, Wang D, Capodanno D, Garg S, Onuma Y, Serruys PW, Gao C; REC-CAGEFREE I Investigators. Drug-Coated Balloon Angioplasty vs Up-Front Stenting for De Novo CAD: 3-Year Follow-Up of REC-CAGEFREE I Trial. J Am Coll Cardiol. 2025 Oct 27:S0735-1097(25)09986-3. doi: 10.1016/j.jacc.2025.10.027. Online ahead of print. PMID 41194754
- [Derived] Gao C, He X, Ouyang F, Zhang Z, Shen G, Wu M, Yang P, Ma L, Yang F, Ji Z, Wang H, Wu Y, Fang Z, Jiang H, Wen S, Liu Y, Li F, Zhou J, Zhu B, Liu Y, Zhang R, Zhang T, Wang P, Liu J, Jiang Z, Xia J, van Geuns RJ, Capodanno D, Garg S, Onuma Y, Wang D, Serruys PW, Tao L; REC-CAGEFREE I Investigators. Drug-coated balloon angioplasty with rescue stenting versus intended stenting for the treatment of patients with de novo coronary artery lesions (REC-CAGEFREE I): an open-label, randomised, non-inferiority trial. Lancet. 2024 Sep 14;404(10457):1040-1050. doi: 10.1016/S0140-6736(24)01594-0. Epub 2024 Sep 2. PMID 39236727
- [Derived] Gao C, He X, Liu Y, Liu J, Jiang Z, Zhu B, Qin X, Xia Y, Zhang T, Wang P, Zhang R, Onuma Y, Xia J, Wang D, Serruys P, Tao L. Drug-coated balloon angioplasty with provisional stenting versus primary stenting for the treatment of de novo coronary artery lesions: REC-CAGEFREE I trial rationale and design. BMC Cardiovasc Disord. 2024 Jun 24;24(1):319. doi: 10.1186/s12872-024-03974-0. PMID 38914951